CLINICAL TRIAL: NCT01539655
Title: A Phase I, Randomized, Open-label, Single-center Study to Assess the Pharmacokinetics of Vandetanib (CAPRELSA) in Healthy Subjects When a Single Oral Dose of Vandetanib 300 mg is Administered Alone and in Combination With Omeprazole or Ranitidine
Brief Title: Study in Healthy Volunteers to Assess Effect of Omeprazole and Ranitidine on the Pharmacokinetics of Vandetanib
Acronym: Vandetanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4200C00101
Record Dates: First submitted 2012-02-10; First posted 2012-02-27 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Medullary Thyroid Cancer
Keywords: Phase 1; healthy volunteers; pharmacokinetics; vandetanib; omeprazole; ranitidine
MeSH Terms: conditions — Carcinoma, Medullary | interventions — vandetanib; Omeprazole; Ranitidine

ARMS (4):
- vandetanib then vandetanib + omeprazole (Experimental): Vandetanib alone in period 1 followed by vandetanib in combination with omeprazole in period 2
  Interventions: Drug: vandetanib; Drug: omeprazole
- vandetanib + omeprazole then vandetanib (Experimental): Vandetanib in combination with omeprazole in period 1 followed by vandetanib alone in period 2
  Interventions: Drug: vandetanib; Drug: omeprazole
- vandetanib then vandetanib + ranitidine (Experimental): Vandetanib alone in period 1 followed by vandetanib in combination with ranitidine in period 2
  Interventions: Drug: vandetanib; Drug: ranitidine
- vandetanib + ranitidine then vandetanib (Experimental): Vandetanib in combination with ranitidine in period 1 followed by vandetanib alone in period 2
  Interventions: Drug: vandetanib; Drug: ranitidine

INTERVENTIONS:
Drug: vandetanib — Oral tablets, 300 mg, single dose
Drug: omeprazole — Oral capsules, 40 mg, multiple doses
  Arms: vandetanib + omeprazole then vandetanib; vandetanib then vandetanib + omeprazole
Drug: ranitidine — Oral tables, 150 mg, multiple doses
  Arms: vandetanib + ranitidine then vandetanib; vandetanib then vandetanib + ranitidine

SUMMARY:
Study in healthy volunteers to assess effect of omeprazole and ranitidine on the pharmacokinetics of vandetanib

DETAILED DESCRIPTION:
A Phase I, Randomized, Open-label, Single-center Study to Assess the Pharmacokinetics of Vandetanib (CAPRELSA) in Healthy Subjects when a Single Oral Dose of Vandetanib 300 mg is Administered Alone and in Combination with Omeprazole or Ranitidine

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures
* Volunteers must be males or females aged 18 to 50 years and with a weight of at least 50 kg and body mass index (BMI) between 18 and 30 kg/m2
* Inclusive Females must have a negative pregnancy test at screening and on admission to the study center
* Females must not be lactating and must be of non childbearing potential defined as postmenopausal or documentation of irreversible surgical sterilization.

Exclusion Criteria:

* History of any clinically significant disease or disorder such as gastrointestinal, hepatic, renal or skin disease.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity
* Volunteers who smoke more than 5 cigarettes per day or are unable to refrain from smoking while resident in the study center
* Screening blood pressure of greater than 140/90 mmHg and/or a resting heart rate of less than 45 beats per minute (repeat test allowed at the Investigator's discretion
* Clinically significant abnormal12-lead ECG as assessed by the Investigator
* QTcF interval greater than 450 ms Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody
* Human immunodeficiency virus (HIV), or positive screen for drugs of abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cmax for a single dose of vandetanib alone and in combination with omeprazole (PPI) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose
AUC(0-t) for a single dose of vandetanib alone and in combination with omeprazole (PPI) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose
Cmax for a single dose of vandetanib alone and in combination with ranitidine (histamine antagonist) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose
AUC(0-t) for a single dose of vandetanib alone and in combination with ranitidine (histamine antagonist) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Treatment period + 7-14 days
ECG data | Treatment period + 7-14 days
Laboratory data | Treatment period + 7-14 days
Vital signs data | Treatment period + 7-14 days
Other PK parameters for a single dose of vandetanib alone and in combination with omeprazole (PPI) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose
Other PK parameters for a single dose of vandetanib alone and in combination with ranitidine (histamine antagonist) | Predose,1,2,3,4,5,6,7,8,10,12,18,24,36,48,72,96,120,144,168,192,216,240,336,504 ,672 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Johansson S, Read J, Oliver S, Steinberg M, Li Y, Lisbon E, Mathews D, Leese PT, Martin P. Pharmacokinetic evaluations of the co-administrations of vandetanib and metformin, digoxin, midazolam, omeprazole or ranitidine. Clin Pharmacokinet. 2014 Sep;53(9):837-47. doi: 10.1007/s40262-014-0161-2. PMID 25117183
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1436&filename=CSR-D4200C00101.pdf
- See also: CSR-D4200C00101.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1436&filename=CSR-D4200C00101.pdf
- See also: Revised_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1436&filename=D4200C00101_Revised_CSP_redacted.pdf